CLINICAL TRIAL: NCT04630561
Title: Great Posture, Great Health - A Community-Based Postural Intervention for Improving Holistic Health
Brief Title: Great Posture, Great Health
Acronym: GPGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin (Ben) D. Holmes, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-004586
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: posture; exercise; community
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects will participate in a 15 minute postural intervention program 2-3 times per week
  Interventions: Behavioral: Postural Intervention Program
- Control Group (No Intervention): Subjects will NOT participate in any postural intervention.

INTERVENTIONS:
Behavioral: Postural Intervention Program — Dynamic warmup program designed to target several areas of physical and mental wellbeing.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to examine the effect of a posture intervention on specific areas of daily function and health: physical, psychological, cognitive, social, and environmental characteristics.

DETAILED DESCRIPTION:
This project promotes community health through postural movement to demonstrate strong physical and mental health benefits. Specifically, Great Posture, Great Health will address two of the top five priorities of general health concerns: 1) obesity and 2) mental health. First, obesity is on the rise although more individuals are meeting or exceeding the current federal physical activity guidelines based on the data provided by the US Department of Health and Human Services (2020). Obesity is a common problem in adults with all socioeconomic status and all races, except Asians. In fact, Asians have low rates of heart disease, asthma, cancer, and a longer life expectancy than other races, potentially due to health behaviors, environment, and stress coping strategies (Acciai et al., 2015). Therefore, we should not overlook the importance of stress coping strategies practiced in Asian countries on obesity. It is becoming more evident that chronic stress (such as elevated cortisol levels) and steroid-based medications are strongly associated with obesity and chronic diseases. It is critical to develop and validate community health strategies to address both priorities. Great Posture, Great Health will introduce one of the most common mind-body postural exercises practiced in Asian countries to a large and diverse population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be physically capable (defined as easy to moderate physical activities daily at least 60 minutes).
* Participants also must have a normal (18.5-24.9kg/m2) or overweight BMI (25-29.9kg/m2).
* Participants must be able to speak, listen, read, and understand sentences written in English.

Exclusion Criteria:

* More than two risk factors for coronary artery disease (high blood pressure, high blood cholesterol level (LDL), family history (a close relative with heart disease), diabetes mellitus, chronic kidney disease
* History of falls, osteoporosis, osteoarthritis, or orthopedic or neurological conditions (i.e., stroke)
* Medications that cause dizziness or slow movement
* Smoke
* Body mass to height squared ratio greater than 30kg/m2 or less than 18.4kg/m2, blood pressure greater than 140/90 mmHg, or a history of heart conditions.
* Individuals with progressive cognitive, neurologic disorders, cancer treatment, chronic heart failure, or unstable medical conditions

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Thigh Strength | 12-week differences (Pre- and Post-intervention measures)
  Isometric measurement (Newtons) of quadriceps and hamstrings musculature
Posture | 12-week differences (Pre- and Post-intervention measures)
  Posture will be measured via the Posture Screen Mobile app. Displacement (mm)
Bone density | 12-week differences (Pre- and Post-intervention measures)
  Bone densiometry will be measured via quantitative ultrasound (Achilles EXPII, GE). T-score.

SECONDARY OUTCOMES:
PROMIS - Physical Activity | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes from a computerized adaptive test (T-score; normative score is 1.0; higher score equates to a better outcome)
PROMIS - Physical Function | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes from a computerized adaptive test (T-score; normative score is 1.0; higher score equates to a better outcome)
PROMIS - Pain Interference | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes from a computerized adaptive test (T-score; normative score is 1.0; higher score equates to a better outcome)
Mindful Attention Awareness Scale (MAAS) | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes (Mean score range: 1-6; higher score equates to increased mindfulness)
Perceived Stress Scale (PSS-10) | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes (Score range: 0-40; higher score equates to increased stress)
Generalized Anxiety Disorder (GAD7) | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes (Score range: 0-21; higher score equates to increased anxiety)
Patient Health Questionnaire Depression Scale (PHQ) | 12-week differences (Pre- and Post-intervention measures)
  Patient Reported Outcomes (Score range: 0-27; score of 10 or greater is considered major depression, 20 or more is severe major depression.)
Sex | Through study completion, an average of 1 year
  Demographic co-variate. (M/F)
Age | Through study completion, an average of 1 year
  Demographic co-variate (years)
BMI | 12-week differences (Pre- and Post-intervention measures)
  Demographic co-variate (BMI index; kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Holmes, DC, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials